CLINICAL TRIAL: NCT05662826
Title: A Virtual Home Intervention to Promote Physical Activity Among Youth With Type 1 Diabetes Part 2
Brief Title: Avatar-based Social Physical Activity
Acronym: ASPA
Status: Suspended | Phase: Not Applicable | Type: Interventional
Why Stopped: Gap in funding
Sponsor: Yale University (Other)
Collaborators: American Heart Association (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2000033736
Record Dates: First submitted 2022-12-14; First posted 2022-12-23 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-08

CONDITIONS: Type 1 Diabetes
Keywords: Exercise; Adolescent; Video games; Self-management; Social support
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Motor Activity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Avatar-based Social Physical Activity (Experimental): Group classes with virtual reality exercise games, talking, acting, and painting activities
  Interventions: Behavioral: Avatar-based Social Physical Activity

INTERVENTIONS:
Behavioral: Avatar-based Social Physical Activity — Exercise, group discussions, role-playing skits, and group painting done in a virtual setting.

SUMMARY:
This study is testing program where teens with type 1 diabetes play Meta Quest 2 virtual reality exercise games and talk, act, and paint about physical activity in virtual meetings with their peers and young adult role models. The outcomes are feasibility and user satisfaction.

ELIGIBILITY:
Inclusion Criteria:

* Age of 14-17 years
* Diagnosis of type 1 diabetes or other absolute insulin deficiency diabetes for ≥6 months
* Moderate-to-vigorous physical activity less than half of recommended levels (defined as ≤3 days per week achieving ≥60min daily MVPA)
* English literacy
* Home Broadband wireless Internet (≥25 mbps downloads, ≥3 mbps uploads on google Internet speed test). This is used in ~98% of US households.
* Willing to use continuous glucose monitor for the duration of participation in the trial.
* Willing to use a computer or smartphone with web camera.
* Under regular care by a healthcare provider (defined as attending at least one appointment in the past year, plus access to verified 24hr phone number to reach the provider's team for insulin dose adjustments if assistance is needed)

Exclusion Criteria:

* A condition or disability besides type 1 diabetes that would preclude participation in group moderate-to-vigorous physical activity (e.g., cerebral palsy, current pregnancy)

Ages: 14 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 24 (Estimated)
Dates: Start 2023-01-17 (Actual); Primary Completion 2026-12-30 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Engagement | 4 weeks
  Number of classes attended
Satisfaction | 4 weeks
  Score on a satisfaction survey that has been custom-designed for the components of this program. Scores range from 0 to 4. A higher score indicates greater satisfaction with the program.

SECONDARY OUTCOMES:
Perceived cohesion | 4 weeks
  Score on perceived cohesion scale (reference 1). Scores range from 0 to 6. A higher score indicates greater cohesion the participant felt among the group.
Motivation for exergame play | 4 weeks
  Score on motivation for exergame play inventory (reference 2). Scores range from 0 to 4. A higher score indicates greater motivation to play the videogame.
Multimodal presence | 4 weeks
  Score on multimodal presence scale (reference 3). Scores range from 0 to 4. A higher score indicates greater feeling of presence in the virtual world.
System usability | 4 weeks
  Score on system usability scale (reference 4). Scores range from 0 to 4. A higher score indicates the system was more feasible to use.

CONTACTS AND LOCATIONS:
Locations (1):
- Yale Children's Diabetes Program, New Haven, Connecticut, United States

IPD SHARING:
Plan to Share IPD: Yes

REFERENCES:
- [Background] Chin WW, Salisbury WD, Pearson AW, Stollak MJ. Perceived cohesion in small groups: Adapting and testing the perceived cohesion scale in a small-group setting. Small Group Research. 1999;30(6):751-766.
- [Background] Staiano, AE, Adams, MA, & Norman, GJ (2019). Motivation for Exergame Play Inventory: Construct validity and relationship to game play. Cyberpsychology: Journal of Psychosocial Research on Cyberspace, 13(3), article 7.
- [Background] Makransky, G., Lilleholt, L., & Aaby, A. (2017). Development and validation of the Multimodal Presence Scale for virtual reality environments: A confirmatory factor analysis and item response theory approach. Computers in Human Behavior, 72, 276-285.
- [Background] Brooke, J. (1996). SUS-A quick and dirty usability scale. Usability evaluation in industry, 189(194), 4-7.